CLINICAL TRIAL: NCT04087928
Title: Efficacy of Focal Muscular Vibration in the Treatment of Upper Limb Spasticity in Subjects With Stroke Outcomes: Randomized Controlled Trial.
Brief Title: Focal Muscular Vibration to Treat Upper Limb Spasticity in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Irene Giovanna Aprile, MD, PhD, Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMV_2019
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Stroke
Keywords: Stroke; Upper limb; Rehabilitation; Focal Muscular Vibration
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Flexors (A) (Experimental): Group A was treated by applying FMV to the flexor muscles of the upper limb (brachial biceps and carpal flexors). Patients will be treated with FMV for three consecutive days: each session consisted of three sessions of 10 minutes each, interspersed with one minute of rest. A vibration frequency of 100 Hz has been applied, according to the literature.
  Interventions: Device: FMV_flex
- Group Extensors (B) (Experimental): Group b was treated by applying FMV to the extensors muscles of the upper limb (triceps brachial and carpus extensors). Patients will be treated with FMV for three consecutive days: each session consisted of three sessions of 10 minutes each, interspersed with one minute of rest. A vibration frequency of 100 Hz has been applied, according to the literature.
  Interventions: Device: FMV_ext

INTERVENTIONS:
Device: FMV_flex — Fisiocomputer EVM (Endomedica, Italy) for application of FMV to flexor muscles of the upper limb (brachial biceps and carpal flexors).
  Arms: Group Flexors (A)
Device: FMV_ext — Fisiocomputer EVM (Endomedica, Italy) for application of FMV to extensors muscles of the upper limb (triceps brachial and carpus extensors).
  Arms: Group Extensors (B)

SUMMARY:
Spasticity following stroke is one of the most debilitating conditions and has a negative influence on the autonomy and quality of life, and greatly worsens the patient's degree of disability. Focal muscular vibration (FMV) is a non-invasive technique to treat spasticity. Has been showed the positive effects of FMV on spasticity in stroke subjects. FMV has been investigated on the antagonist muscle, as well as directly on the spastic muscle, showing in both cases a significant reduction in spasticity. However, isn't unclear which is the most effective in the treatment of spasticity.

The objective of the study is to evaluate the efficacy of FMV of the muscles of the upper limb in subjects with subacute stroke, comparing the effects obtained by treating the spastic muscles directly versus to those obtained by treating the respective antagonist muscles.

DETAILED DESCRIPTION:
Stroke is the major cause of permanent disability with an incidence in Italy of 293 affected persons per 100,000 inhabitants. The onset of spasticity following stroke (20-46%) is one of the most disabling conditions and has a negative influence on the patient's autonomy and quality of life.

The development of spasticity during the rehabilitation process of these patients is a very limiting factor for the functional recovery of the affected side. The onset of spasticity considerably worsens the patient's degree of disability.

Focal muscular vibration (FMV) is a non-invasive technique to treat spasticity. Has been showed the positive effects of FMV on spasticity in stroke subjects.

Introduced by Hagbarth and Eklund at the end of the 1960s, it is based on the tonic-vibratory reflex. Based on this mechanism, some authors suggest that the FMV should be applied to the antagonist muscle in order to obtain a significant reduction in spasticity. However the literature shows a reduction in spasticity through the application of FMV directly on the spastic muscle. These effects seem to be related to the stimulation of cortical motor areas. Nevertheless, it remains unclear which approach is most effective in treating of spasticity.

Stroke is a very common pathology, as well as a rehabilitative and social problem which also affects welfare. Considering prevalence of spasticity in stroke patients and the effects on their functional recovery, it is important to identify the most effective treatment to guarantee a more suitable rehabilitation process. In addition to this, it is worth remembering that FMV is less invasive and has lower costs than botulinum toxin, the current gold standard in the treatment of spasticity.

The objective of the study is to evaluate the efficacy of FMV of the muscles of the upper limb in subjects with subacute stroke, comparing the effects obtained by treating the spastic muscles directly versus to those obtained by treating the respective antagonist muscles. Specifically, the two approaches will be compared on: (i) the reduction of the degree of spasticity, assessed by clinical scales and with an instrumental protocol; (ii) motor performance of the patient, using a robotic system; (iii) pain reduction.

ELIGIBILITY:
Inclusion Criteria:

* first cerebral stroke
* 2 weeks up to 12 months post the acute event (subacute patients)
* age between 35-80 years
* single cortical or subcortical event
* spastic paresis of the upper limb (Modified Ashworth Scale score ≥ 2)
* ability to give written consent
* compliance with the study procedures

Exclusion Criteria:

* comorbidities affecting the paretic upper limb (fractures, trauma or peripheral neuropathies)
* cognitive and/or communicative disability (e.g. due to brain injury): inability to understand the instructions required for the study
* treatment with focal or systemic antispastic drugs (i.e. baclofen, thiocolchicoside, tizanidine).

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Change in Modified Ashworth Scale (MAS) | Baseline (T0), Treatment (1 weeks) (T1), Follow up (4 weeks ) (T2)
  The MAS is a 6 point ordinal scale used for grading hypertonia in individuals with neurological diagnoses. A score of 0 on the scale indicates no increase in tone while a score of 4 indicates rigidity. Tone is scored by passively moving the individual's limb and assessing the amount of resistance to movement felt by the examiner.

SECONDARY OUTCOMES:
Change in Motricity Index (MI) | Baseline (T0), Treatment (1 weeks) (T1), Follow up (4 weeks ) (T2)
  The MI aims to evaluate lower limb motor impairment after stroke, administrated on both sides.
  Items to assess the lower limbs are 3, scoring from 0 to 33 each: (1) ankle dorsiflexion with foot in a plantar flexedposition (2) knee extension with the foot unsupported and the knee at 90° (3) hip flexion with the hip at 90° moving the knee as close as possible to the chin. (no movement: 0, palpable flicker but no movement: 9, movement but not against gravity :14, movement against gravity movement against gravity: 19, movement against resistance: 25, normal:33).
Change in ID Pain | Baseline (T0), Treatment (1 weeks) (T1), Follow up (4 weeks ) (T2)
  The ID Pain questionnaire (ID-P) is used to evaluate presence of neuropathic pain. Is a tool composed of a six dichotomous answer questions (yes/no). The total score is calculated by assigning a point for each 'yes' to question 1-5 and no points for every 'no'. Instead, a point is subtracted for 'yes' to question 6 and no points are assigned for 'no'. A score equal to greater than '3' indicates a presence of neuropathic pain.
Change in Neuropathic Pain four Questions (DN4) | Baseline (T0), Treatment (1 weeks) (T1), Follow up (4 weeks ) (T2)
  The DN4 used to evaluate presence of neuropathic pain, and consist of a brief interview of four questions answered yes/no: two on what the patient has conceived and two during the exam for the evaluation of hypoesthesia to the touch or sting and the evaluation of allodynia with the skimming of the skin. For each 'yes' a point is assigned. The total score is given by the sum of the individuals. The cut off for the presence of neuropathic pain is '4'.
Change in Neuropathic Pain Symptom Inventory (NPSI) | Baseline (T0), Treatment (1 weeks) (T1), Follow up (4 weeks ) (T2)
  The NPSI consist of ten descriptors of neuropathic pain plus two elements for the duration of spontaneous and paroxysmal pains. The tool evaluates mean pain intensity in the last 24h in a verbal numeric scale from zero (no pain) to 10 (worst imaginable pain). Total pain intensity score may be calculated by the sum of 10 descriptors.
Change in Numerical Rating Scale (NRS) | Baseline (T0), Treatment (1 weeks) (T1), Follow up (4 weeks ) (T2)
  The NRS is a quantitative one-dimensional numerical scale of pain assessment at 11 points; the scale requires the operator to ask the patient to select the number that best describes the intensity of hi s pain, from 0 to 10, at that precise moment.

OTHER OUTCOMES:
Reaching movements | Baseline (T0), Treatment (1 weeks) (T1), Follow up (4 weeks ) (T2)
  Reaching movements are evaluated by the robot Motore (Humanware).
Tone of the fingers | Baseline (T0), Treatment (1 weeks) (T1), Follow up (4 weeks ) (T2)
  Assessment of the finger tone, measured in Newton (N), is obtained through Amadeo (Tyromotion).
Strength of the fingers | Baseline (T0), Treatment (1 weeks) (T1), Follow up (4 weeks ) (T2)
  Assessment of the finger strength, measured in Newton (N), is obtained through Amadeo (Tyromotion).

CONTACTS AND LOCATIONS:
Overall Officials: Irene Aprile, MD, PhD, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi
Locations (1):
- Irene Aprile, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Murillo N, Valls-Sole J, Vidal J, Opisso E, Medina J, Kumru H. Focal vibration in neurorehabilitation. Eur J Phys Rehabil Med. 2014 Apr;50(2):231-42. PMID 24842220
- [Result] Hagbarth KE, Eklund G. Tonic vibration reflexes (TVR) in spasticity. Brain Res. 1966 Aug;2(2):201-3. doi: 10.1016/0006-8993(66)90029-1. No abstract available. PMID 5968925
- [Result] Ageranoti SA, Hayes KC. Effects of vibration on hypertonia and hyperreflexia in the wrist joint of patients with spastic hemiparesis. Physiotherapy Canada 1990;42:24-33.
- [Result] Liepert J, Binder C. Vibration-induced effects in stroke patients with spastic hemiparesis--a pilot study. Restor Neurol Neurosci. 2010;28(6):729-35. doi: 10.3233/RNN-2010-0541. PMID 21209488
- [Result] Noma T, Matsumoto S, Shimodozono M, Etoh S, Kawahira K. Anti-spastic effects of the direct application of vibratory stimuli to the spastic muscles of hemiplegic limbs in post-stroke patients: a proof-of-principle study. J Rehabil Med. 2012 Apr;44(4):325-30. doi: 10.2340/16501977-0946. PMID 22402727
- [Result] Caliandro P, Celletti C, Padua L, Minciotti I, Russo G, Granata G, La Torre G, Granieri E, Camerota F. Focal muscle vibration in the treatment of upper limb spasticity: a pilot randomized controlled trial in patients with chronic stroke. Arch Phys Med Rehabil. 2012 Sep;93(9):1656-61. doi: 10.1016/j.apmr.2012.04.002. Epub 2012 Apr 13. PMID 22507444
- [Result] Shaw L, Rodgers H, Price C, van Wijck F, Shackley P, Steen N, Barnes M, Ford G, Graham L; BoTULS investigators. BoTULS: a multicentre randomised controlled trial to evaluate the clinical effectiveness and cost-effectiveness of treating upper limb spasticity due to stroke with botulinum toxin type A. Health Technol Assess. 2010 May;14(26):1-113, iii-iv. doi: 10.3310/hta14260. PMID 20515600
- [Result] Aprile I, Di Sipio E, Germanotta M, Simbolotti C, Padua L. Muscle focal vibration in healthy subjects: evaluation of the effects on upper limb motor performance measured using a robotic device. Eur J Appl Physiol. 2016 Apr;116(4):729-37. doi: 10.1007/s00421-016-3330-1. Epub 2016 Jan 27. PMID 26818756